CLINICAL TRIAL: NCT03282682
Title: Strength Training as a Supplemental Therapy of Androgen Deficiency of the Aging Male (ADAM)
Brief Title: Strength Training as a Supplemental Therapy of Androgen Deficiency of the Aging Male
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Comenius University (Other)
Collaborators: Norwegian School of Sport Sciences (Other); Slovak Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Milan Sedliak, Independent researcher, Vice-dean for science, research and international cooperation, Comenius University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FSPORT-CU-ADAM
Record Dates: First submitted 2017-08-20; First posted 2017-09-14 (Actual); Results first posted 2020-05-05 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Hypogonadism, Male; Physical Activity; Testosterone Deficiency
Keywords: hypogonadism; aging male; strength training; physical activity; testosterone
MeSH Terms: conditions — Eunuchism; Motor Activity; Hypogonadism | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: The study is 3 arms 12-week strength training program to assess the effect of testosterone replacement therapy (TRT) with strength training (ST) and strength training (ST) for hypogonadal patients without testosterone replacement therapy (NON-TRT) with control healthy eugonadal group, that is also engaged in strength training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- hypogonadal males without TRT (Experimental): Strength training
  Interventions: Procedure: Strength training
- hypogonadal males with TRT (Experimental): Strength training and regular prescribed testosterone therapy given by participant urologist.
  Interventions: Procedure: Strength training
- healthy eugonadal males (Active Comparator): Strength training
  Interventions: Procedure: Strength training

INTERVENTIONS:
Procedure: Strength training — The participants perform strength training sessions two times per week for 12 weeks. Each training session include 5-minute general dynamic warm-up followed by progressive strength training with exercises for the entire body. The strength exercises are performed with free weights and on machines. The training program consist of 6 exercises for upper and lower body at an intensity of 60-80% (8 - 12RM: the load that induces technique failure in eight or twelve repetitions) of one-repetition maximum and takes approximately 60 minutes. The exercises performed are: leg press, split squats, bench press, knee extension, knee flexion, seated cable rows, seated cable pull downs, dumbbell bench press, incline dumbbell bench press.

SUMMARY:
This study examines the effect of 12-week strength training program with and without testosterone replacement therapy (TRT) on body composition, physical function, selected biochemical markers of metabolic health, molecular parameters of training adaptation and the quality of life patients with ADAM. The investigators believe, that strength training program performed 2 times per week for 12 weeks can improve body composition (decrease fat mass and gain lean mass), muscle strength, muscle power and general quality of life in all training groups. In addition, combination TRT and strength training could help decrease fat mass, improve BMI, cardio-respiratory fitness and thus provide optimal therapy combination for hypogonadal ageing males.

DETAILED DESCRIPTION:
The study is 3 groups controlled 12-week study to assess the effect of testosterone replacement therapy (TRT) with strength training (ST) and strength training (ST) for hypogonadal participants without testosterone replacement therapy (NON-TRT) with control healthy eugonadal group, that is also engaged in strength training.

Strength training protocol starts one week after all the pre-intervention testing. The intervention is performed at the Comenius University in Bratislava, Faculty of Physical Education and Sport (FSPORT CU) in Slovakia. The strength training protocol follows a modified resistance exercise program. The participants perform strength training sessions two times per week for 12 weeks. All training sessions are supervised and guided by professional coaches with university degree in sports training to ensure safety, technique and progression in training load, with a maximum of three participants per coach.

Each training session include 5-minute general dynamic warm-up followed by progressive strength training with exercises for the entire body. The strength exercises are performed with free weights and on machines. The training program consist of 6 exercises for upper and lower body at an intensity of 60-80% (8 - 12RM: the load that induces technique failure in eight or twelve repetitions) of one-repetition maximum and takes approximately 60 minutes. The participants are instructed to perform concentric action in 2 s and immediately after eccentric action in also 2 s. The exercises performed are: leg press, split squats, bench press, knee extension, knee flexion, seated cable rows, seated cable pull downs, dumbbell bench press, incline dumbbell bench press. Training equipment is provided by KOHI Leopoldov, Slovakia and Technogym, Italia.

Clinical and muscle cellular outcomes are collected before the intervention (pre-testing assessments) and after the intervention (post-testing assessments). Post intervention measurements start 7 days after intervention and go up to 3 weeks after intervention.

Clinical outcomes Body composition analysis is measured by Dual-energy X-ray Absorptiometry using Hologic fan-beam bone densitometer Discovery QDR series. LBM(lean body mass) is measured in total body and separately for arms, legs and trunk. The changes in lower and upper body LBM are investigated separately because of differences in androgen sensitivity in leg muscles compared to neck, chest and shoulder muscles. Body weight is measured by bioimpedance scale, the height by stadiometer and waist circumference by tape. The body mass index is calculated.

Biochemical outcomes Fasting morning venous blood is taken from 8:00 am to 10:00 am. The haematological and biochemical parameters analysed are Haemoglobin, hematocrits, leucocytes, thrombocytes, glucose, urea, sodium, potassium, calcium, ALAT, total cholesterol, LDL cholesterol, HDL cholesterol, triglyceride, testosterone, oestrogen, LH, FSH, SHBG, albumin, bilirubin, total protein, CRP, insulin, PSA.

Physical functioning Muscle strength is measured by novel portable isometric knee dynamometer (maximal voluntary contraction of isometric knee extension, isometric knee flexion), hand grip strength dynamometry by Camry Digital Hand Dynamometer, predicted 1RM leg press from multiple repetition maximum testing. Cardio-respiratory fitness is measured by The Single Stage Treadmill Walking Test on Woodway Pro Treadmill, 10-m fast walk and 10-m usual walk measured by Photocells.

Quality of life The general health status is measured by The Short Form (36) Health Survey patient-reported survey of patient health (SF-36). In addition to that clinically investigating the health-related quality of life (HRQoL) and symptoms of aging men are measured by Aging Males' Symptom Scale (AMS).

Muscle cellular outcomes Muscle biopsies are obtain from approximately 80% of the subjects included in the study. Participants not willing to undergo biopsy are still eligible for trial participation.

With the participant in a supine position, a 5 mm Muscle Biopsy Cannula (Bergstrom-stille, Sweden) with manual suction is used to obtain muscle samples (200 mg), under local anaesthesia (Lidocain 2%,). Before the intervention the biopsy is obtained from the mid-section of the right musculus vastus lateralis, and after the intervention the biopsy is obtained 3 cm proximal to the pre-intervention biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients of secondary hypogonadism on testosterone replacement therapy, newly diagnosed patients of secondary hypogonadism.

Exclusion Criteria:

* Regular strength training, medical treating osteoporosis, abnormal digital rectal results, conditions which are medical contraindications (without adjusting state): diabetes mellitus, severe cardiac arrhythmia, uncontrolled hypertension, unstable angina pectoris, chronic obstructive pulmonary disease, epilepsy, unstable bone lesions with high risk of fracture, prostate cancer or abnormal serum PSA levels without adverse histological examination.

Ages: 45 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milan Sedliak, assoc. prof., Principal Investigator — Comenius University of Bratislava, Faculty Physical Education and Sport
Locations (1):
- Comenius University in Bratislava, Faculty of physical education and sport, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Basaria S. Androgen deprivation therapy, insulin resistance, and cardiovascular mortality: an inconvenient truth. J Androl. 2008 Sep-Oct;29(5):534-9. doi: 10.2164/jandrol.108.005454. Epub 2008 Jun 20. PMID 18567642
- [Result] Hildreth KL, Barry DW, Moreau KL, Vande Griend J, Meacham RB, Nakamura T, Wolfe P, Kohrt WM, Ruscin JM, Kittelson J, Cress ME, Ballard R, Schwartz RS. Effects of testosterone and progressive resistance exercise in healthy, highly functioning older men with low-normal testosterone levels. J Clin Endocrinol Metab. 2013 May;98(5):1891-900. doi: 10.1210/jc.2013-2227. Epub 2013 Mar 26. PMID 23533227
- [Result] Schwarz ER, Willix RD Jr. Impact of a physician-supervised exercise-nutrition program with testosterone substitution in partial androgen-deficient middle-aged obese men. J Geriatr Cardiol. 2011 Dec;8(4):201-6. doi: 10.3724/SP.J.1263.2011.00201. PMID 22783306
- [Result] Kadi F, Bonnerud P, Eriksson A, Thornell LE. The expression of androgen receptors in human neck and limb muscles: effects of training and self-administration of androgenic-anabolic steroids. Histochem Cell Biol. 2000 Jan;113(1):25-9. doi: 10.1007/s004180050003. PMID 10664066
- [Result] Gardner JR, Livingston PM, Fraser SF. Effects of exercise on treatment-related adverse effects for patients with prostate cancer receiving androgen-deprivation therapy: a systematic review. J Clin Oncol. 2014 Feb 1;32(4):335-46. doi: 10.1200/JCO.2013.49.5523. Epub 2013 Dec 16. PMID 24344218
- [Derived] Kralik M, Cvecka J, Buzgo G, Putala M, Ukropcova B, Ukropec J, Killinger Z, Payer J, Kollarik B, Bujdak P, Raastad T, Sedliak M. Strength training as a supplemental therapy for androgen deficiency of the aging male (ADAM): study protocol for a three-arm clinical trial. BMJ Open. 2019 Sep 5;9(9):e025991. doi: 10.1136/bmjopen-2018-025991. PMID 31492775

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hypogonadal Males Without TRT | Hypogonadal Males With TRT | Healthy Eugonadal Males
Started | 6 | 8 | 8
Completed | 6 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypogonadal Males Without TRT | Hypogonadal Males With TRT | Healthy Eugonadal Males | Total
Number analyzed (Participants) | 6 | 8 | 8 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.41 (7.9) | 43.03 (2.9) | 50.11 (5.1) | 47.07 (7.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 6 | 8 | 8 | 22
Race/Ethnicity, Customized [Number; unit: participants]
  Slovak | 6 | 8 | 8 | 22
Region of Enrollment [Number; unit: participants]
  Slovakia | 6 | 8 | 8 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Lean Mass
Description: Total body by Dual-energy X-ray Absorptiometry using Hologic fan-beam bone densitometer Discovery QDR series.
Time Frame: 7 days before intervention, 7 days after intervention
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Hypogonadal Males Without TRT | Hypogonadal Males With TRT | Healthy Eugonadal Males
Number analyzed (Participants) | 6 | 8 | 8
grams | 2734 (1967) | 499 (1566) | 2268 (2609)

2. Secondary Outcome: Change From Baseline in Fat Mass
Description: Total body by Dual-energy X-ray Absorptiometry using Hologic fan-beam bone densitometer Discovery QDR series.
Time Frame: 7 days before intervention, 7 days after intervention
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Hypogonadal Males Without TRT | Hypogonadal Males With TRT | Healthy Eugonadal Males
Number analyzed (Participants) | 6 | 8 | 8
grams | -1969 (2526) | -1263 (1920) | -755 (1514)

3. Secondary Outcome: Change From Baseline in Total Body Mass
Description: Total body by Dual-energy X-ray Absorptiometry using Hologic fan-beam bone densitometer Discovery QDR series.
Time Frame: 7 days before intervention, 7 days after intervention
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Hypogonadal Males Without TRT | Hypogonadal Males With TRT | Healthy Eugonadal Males
Number analyzed (Participants) | 6 | 8 | 8
grams | 621.53 (2922.45) | -821.73 (3279.29) | 1435.04 (3655.01)

4. Secondary Outcome: Change From Baseline in 10-m Usual Walk Test
Description: Measured in seconds by Microgates Photocells and than calculated to meters per second.
Time Frame: 7 days before intervention, 7 days after intervention
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Hypogonadal Males Without TRT | Hypogonadal Males With TRT | Healthy Eugonadal Males
Number analyzed (Participants) | 6 | 8 | 8
m/s | 0 (0.089) | -0.06 (0.146) | -0.05 (0.136)

5. Secondary Outcome: Change From Baseline in 10-m Fast Walk Test
Description: Measured in seconds by Microgates Photocells than calculated to meters per second
Time Frame: 7 days before intervention, 7 days after intervention
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Hypogonadal Males Without TRT | Hypogonadal Males With TRT | Healthy Eugonadal Males
Number analyzed (Participants) | 6 | 8 | 8
m/s | 0.05 (0.255) | -0.1 (0.172) | -0.13 (0.253)

6. Secondary Outcome: Change From Baseline in Handgrip Strength
Description: Measured by Camry Digital Hand Dynamometer.
Time Frame: 7 days before intervention, 7 days after intervention
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Hypogonadal Males Without TRT | Hypogonadal Males With TRT | Healthy Eugonadal Males
Number analyzed (Participants) | 6 | 8 | 8
kg | -1.41 (4.00) | 0.84 (2.12) | -0.02 (3.28)

7. Secondary Outcome: Change From Baseline in Maximal Voluntary Contraction (MVC) of Isometric Knee Extension
Description: Measured by Portable Isometric Knee Dynamometer.
Time Frame: 7 days before intervention, 7 days after intervention
Measure: Mean (Standard Deviation); unit: Nm
Arm/Group | Hypogonadal Males Without TRT | Hypogonadal Males With TRT | Healthy Eugonadal Males
Number analyzed (Participants) | 6 | 8 | 8
Nm | -9.65 (93.44) | 8.15 (28.97) | 1.35 (69.50)

8. Secondary Outcome: Change From Baseline in Maximal Voluntary Contraction (MVC) of Isometric Knee Flexion
Description: Measured by Portable Isometric Knee Dynamometer.
Time Frame: 7 days before intervention, 7 days after intervention
Measure: Mean (Standard Deviation); unit: Nm
Arm/Group | Hypogonadal Males Without TRT | Hypogonadal Males With TRT | Healthy Eugonadal Males
Number analyzed (Participants) | 6 | 8 | 8
Nm | 2.32 (27.89) | 24.64 (36.09) | 14.36 (28.13)

9. Secondary Outcome: Change From Baseline in The Single Stage Treadmill Walking Test
Description: This test is focused on calculated VO2max in ml.kg-1.min-1 from speed measured on Woodway Pro Treadmill.
Time Frame: 7 days before intervention, 7 days after intervention
Measure: Mean (Standard Deviation); unit: ml.kg-1.min-1
Arm/Group | Hypogonadal Males Without TRT | Hypogonadal Males With TRT | Healthy Eugonadal Males
Number analyzed (Participants) | 6 | 8 | 8
ml.kg-1.min-1 | 0.61 (0.64) | 0.25 (0.64) | 0.42 (0.54)

10. Secondary Outcome: Change From Baseline in Predicted One Repetition Maximum on Leg Press
Description: One repetition maximum in kg on leg press is predicted from multiple repetition maximum testing and measured on Life Fitness Signature Series Leg Press machine.
Time Frame: 7 days before intervention, 7 days after intervention
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Hypogonadal Males Without TRT | Hypogonadal Males With TRT | Healthy Eugonadal Males
Number analyzed (Participants) | 6 | 8 | 8
kg | 45.31 (28.39) | 51.59 (34.43) | 51.40 (27.16)

11. Secondary Outcome: Change From Baseline in Maximal Voluntary Contraction in Benchpress
Description: Measured in N by FiTRO Force Plates.
Time Frame: 7 days before intervention, 7 days after intervention
Measure: Mean (Standard Deviation); unit: N
Arm/Group | Hypogonadal Males Without TRT | Hypogonadal Males With TRT | Healthy Eugonadal Males
Number analyzed (Participants) | 6 | 8 | 8
N | -6.49 (147.12) | 64.31 (143.29) | 66.68 (103.38)

12. Secondary Outcome: Change From Baseline in The Short Form Health Survey (SF-36)
Description: Patient-reported survey of patient health (SF-36), clinically investigating the health-related quality of life (HRQoL). The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. The items contributing to a scale are scored so that a higher score represents better health, and they are averaged together to create the scale score.
Time Frame: 7 days before intervention, 7 days after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hypogonadal Males Without TRT | Hypogonadal Males With TRT | Healthy Eugonadal Males
Number analyzed (Participants) | 6 | 8 | 8
score on a scale | 2.50 (9.87) | 7.50 (18.52) | 3.75 (12.46)

13. Secondary Outcome: Change From Baseline in Aging Males' Symptom (AMS) Scale
Description: Measuring symptoms of ageing men by numeric score scale.
  The questionnaire has for each of the 17 item an option to check one of 5 degrees of severity (severity 1...5 points at the questionnaire).
  The composite scores for each of the three dimensions (sub-scales) is based on adding up the scores of the items of the respective dimensions. The composite score (total score) is the sum of the three dimension scores. Higher score means higher severity of symptoms. The minimum total score is 17 and the maximum is 85.
Time Frame: 7 days before intervention, 7 days after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hypogonadal Males Without TRT | Hypogonadal Males With TRT | Healthy Eugonadal Males
Number analyzed (Participants) | 6 | 8 | 8
score on a scale | -4.83 (7.41) | -2.00 (5.98) | -6.25 (5.09)

14. Secondary Outcome: Change From Baseline in Metabolic Parameters
Description: Fasting morning venous blood was taken after overnight (10-hour) fasting and 15 min rest from cubital vein from 8:00 am to 10:00 am [69] into closed system collection tubes containing beads coated with a clotting activator and polyacryl ester-gel (Sarstedt AG & Co, Germany). The blood will be centrifuged (3000g, 4°C, 10min) immediately after sampling to obtain EDTA plasma or they will be centrifuged (3000g, 4°C, 20min) after 30min at RT, to obtain serum.
Time Frame: 7 days before intervention, 7 days after intervention
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Hypogonadal Males Without TRT | Hypogonadal Males With TRT | Healthy Eugonadal Males
Number analyzed (Participants) | 6 | 8 | 8
mmol/l
  S-Bilirubin | 0.0006 (0.0038) | 0.0008 (0.004) | -0.003 (0.006)
  S-Creatinine | -0.006 (0.008) | -0.0002 (0.0052) | 0.0011 (0.0038)
  S-Glucose | 0.33 (0.44) | 0.29 (0.50) | -0.02 (0.65)
  S-Total Cholesterol | 0.10 (0.67) | 0.22 (0.71) | 0.29 (1.11)
  S-HDL Cholesterol | 0.06 (0.10) | 0.09 (0.17) | 0.08 (0.20)
  S-LDL Cholesterol | -0.06 (0.52) | -0.30 (1.07) | -0.12 (0.84)
  S-Triglyceride | -0.20 (0.46) | 0.38 (1.27) | 0.28 (0.86)
  S-Urea | -0.16 (1.45) | 3.77 (8.58) | 0.84 (1.26)
  S-Uric Acid | -0.016 (0.071) | 0.004 (0.047) | -0.010 (0.053)

15. Secondary Outcome: Change From Baseline in Liver Function Blood Parameters
Description: as for outcome 14
Time Frame: 7 days before intervention, 14 days after intervention
Measure: Mean (Standard Deviation); unit: µkat/l
Arm/Group | Hypogonadal Males Without TRT | Hypogonadal Males With TRT | Healthy Eugonadal Males
Number analyzed (Participants) | 6 | 8 | 8
µkat/l
  S-ALP | 0.06 (0.11) | 0.05 (0.11) | 0.10 (0.18)
  S-ALT | 0.19 (0.49) | -0.05 (0.28) | -0.07 (0.10)
  S-AMS | 0.06 (0.23) | 0.05 (0.08) | 0.07 (0.16)
  S-AST | 0.05 (0.19) | 0.00 (0.19) | -0.01 (0.04)
  S-GMT | -0.13 (0.23) | 0.01 (0.16) | -0.05 (0.27)

16. Secondary Outcome: Change From Baseline in Hormonal Parameters
Description: as for outcome 14
Time Frame: 7 days before intervention, 14 days after intervention
Measure: Mean (Standard Deviation); unit: nmol/l
Arm/Group | Hypogonadal Males Without TRT | Hypogonadal Males With TRT | Healthy Eugonadal Males
Number analyzed (Participants) | 6 | 8 | 8
nmol/l
  S-Testosterone | 1.69 (1.20) | -0.50 (3.51) | -1.99 (2.59)
  S-SHBG | 2.42 (4.67) | -1.35 (6.10) | -2.93 (6.55)
  S-Cortisol | -32.93 (103.28) | -44.60 (140.83) | 34.34 (159.29)
  S-Insuline | 0.004 (0.046) | 0.019 (0.061) | 0.006 (0.023)

17. Secondary Outcome: Change From Baseline in Ions
Description: as for outcome 14
Time Frame: 7 days before intervention, 14 days after intervention
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Hypogonadal Males Without TRT | Hypogonadal Males With TRT | Healthy Eugonadal Males
Number analyzed (Participants) | 6 | 8 | 8
mmol/l
  S-Chlorides | -1.47 (2.50) | -0.77 (4.21) | -0.33 (3.78)
  S-Potassium | 0.17 (0.34) | 0.06 (0.13) | 0.14 (0.31)
  S-Sodium | 0.08 (1.26) | -0.15 (1.31) | -0.19 (1.13)

18. Secondary Outcome: Change From Baseline in CRP
Description: as for outcome 14
Time Frame: 7 days before intervention, 14 days after intervention
Measure: Mean (Standard Deviation); unit: mg/l
Arm/Group | Hypogonadal Males Without TRT | Hypogonadal Males With TRT | Healthy Eugonadal Males
Number analyzed (Participants) | 6 | 8 | 8
mg/l | 0.02 (9.40) | 0.13 (2.26) | -1.67 (2.40)

19. Secondary Outcome: Change From Baseline in Muscle Fiber Size
Description: Muscle fiber size measured in um2. Analysis of the date are in progress.
Time Frame: 7 days before intervention, 14 days after intervention
Reporting Status: Not Posted, anticipated posting 2021-12

20. Secondary Outcome: Change From Baseline in Regulators of Muscle Fiber Size
Description: Regulators of muscle fiber size - number of myonuclei per muscle fiber, number of satellite cells per muscle fiber, number of satellite cells and myonuclei positive for androgen receptors, proteins involved in muscle hypertrophy. Analysis of the date are in progress.
Time Frame: 7 days before intervention, 14 days after intervention
Reporting Status: Not Posted, anticipated posting 2021-12

ADVERSE EVENTS:
Time Frame: 3 months
Description: This type of supervised exercise interventions are very well-tolerated and no major risks and all-cause mortalities are expected. The intervention protocol was also well-tolerated, well-attended, with exercise session attendance approximately 90%, without any serious adverse events during the intervention, when supervised and controlled by specialists trained in this field.
Arm/Group | Hypogonadal Males Without TRT | Hypogonadal Males With TRT | Healthy Eugonadal Males
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
The major limit of the study was low number of the newly diagnosed patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT03282682/Prot_SAP_000.pdf